#### PROTOCOL TITLE:

Improving Employment and Reducing Recidivism among Prison Offenders via Virtual Interview Training Tool

#### PRINCIPAL INVESTIGATOR:

Name: Matthew J. Smith, PhD, MSW, MPE, LCSW

Department: School of Social Work Telephone Number: (734) 764-3309 Email Address: mattjsmi@umich.edu

**VERSION DATE: June 11, 2020** 

**CLINICALTRIALS:** NCT04140942

### Modifying and Evaluating Virtual Interview Training for Villagers

Consent to participate in a Research Study

### **Principal Investigator:**

Matthew J. Smith, Ph.D., School of Social Work, University of Michigan

### Invitation to Participate in a Research Study

We invite you to be part of a research study to test if a new computer program improves job interviewing skills. We are asking you to be part of this study because:

- 1) You are at least 36 years old
- 2) You are living in a Vocational Village that is participating in this study
- 3) You are within 3 months of your earliest release date

# Important Information about the Research Study

Villagers may have difficulty finding jobs. A virtual reality app was created to try to improve interviewing skills for villagers transitioning back into society. We are asking you to be part of a research study. We want to test the virtual reality app to see if it helps improve interview skills and helps villagers find jobs.

The Virtual Reality Job Interview Training (VR-JIT) tool, also known as 'Molly' who is your virtual interviewer, will allow you practice interviewing with a virtual human resource staff who is looking to hire someone for their department store. Vocational Village staff will help you learn how to use this tool and practice some job interviews. Your goal will be to successfully interview and obtain the virtual job. The goal is to help you gain better job interview skills.

This study is funded by the Michigan Institute for Clinical and Health Research (MICHR) at the University of Michigan.

#### **Description of Your Involvement**

#### If you join this study:

Villagers will be randomly assigned (like the flip of a coin) to one of the two conditions.

**Group 1:** Participants will get the usual job interview training provided through the Vocational Village.

**Group 2:** Participants will get the usual job interview training provided through the Vocational Village as well as job interview training using the Molly training.

#### **Study Visits:**

The research study will take place over a series of visits. At the first few visits you will meet with UM research staff to complete some surveys about your background and life stress. You will also complete a practice job interview role play that will be audio and video recorded. Then, you complete some more surveys and questionnaires. You will then be randomly assigned to Condition 1 or Condition 2.

If you are assigned to Condition 1, you will participate in job interview training provided through the Vocational Village as usual. This will include normal class-time procedures, job skill training, and mock interviewing.

If you are assigned to Condition 2, you will be trained to use the Molly training along with the usual job interview training provided by the Vocational Village. You will then be asked to complete practice job interviews using this program for approximately 4-6 weeks. Each interview lasts approximately 30 minutes. You will have general access to the tool.

After you have completed approximately 15 interviews using the Molly training, study staff will conduct another study visit with you. You will again complete some surveys, a practice job interview role play with study staff that will be audio and video recorded, and other survey measures. If you are assigned to Condition 2, you will also be asked to complete some surveys on your acceptability and usability of the Molly training.

You will also complete a 6-month and 12-month follow up survey. The follow up survey will be approximately 10-15 minutes and will measure your current employment status and life stress. We will obtain your contact information from MDOC in order to reach you. If we are unable to reach you, we will ask MDOC to let us know whether or not you are currently employed. For all participants, MDOC will share with us if you are currently released or incarcerated as well as if you are still a Vocational Villager.

#### **Benefits of Participation**

Since the training was created to improve the ability to interview, you may receive some direct benefit from participating. We hope that what we find out in this study will help us to create better interview training for other villagers. There are no direct benefits for the villagers assigned to Condition 1 during data collection, however, these villagers will gain access to the tool once all their study data has been collected.

### Risks and Discomforts of Participation

There is a rare confidentiality risk that the University of Michigan computer server system could be breached or that your identity will be compromised. We will reduce this risk by storing your data on the server protected by passwords and a firewall.

Spending 45 minutes using the tool could cause fatigue or boredom. Please let someone know if you need a break. Also, we will offer you a 5-minute break during the in-person study visits.

You may become upset due to the sensitive nature of the questions. You will be allowed to skip any questions you do not want to answer.

There is a risk that someone outside of the study team, including prison personnel, may attempt to access the data. However, all effort will be made to prevent this. All surveys will only have PINs, so even if Vocational Village staff somehow sees completed surveys or forms, they will be unable to identify who completed them. Vocational Village staff will not collect or view any of the survey information collected by study participants during the first visits.

The Vocational Village staff may overhear your interaction with the Molly training.

## Incentive to be in the Study

You will receive \$40 in gift cards for completing the two follow up surveys after your release. You will receive one \$20 gift card after completion of the 6-month follow up survey and one \$20 gift card after completion of the 12-month follow up survey. Therefore, you can receive up to \$40 for your participation.

#### Confidentiality

We will not include any information that would identify you. We will protect your privacy by completing all research visits in a private or semi-private research room. There may be Vocational Village cameras in the room in which you use the tool, as well as in the semi-private room where you will be interviewed. MDOC will also know who participated in this study. To keep your information safe, the researchers will enter study data on a computer that is protected by a password. To protect your confidentiality, your name will not be in any written or published materials. All information will only be used for research and statistical purposes and data will not be shared with correctional officials. The researchers will keep this information indefinitely for future research about virtual reality interventions.

The video and audio recordings from the mock interviews will be taken out of the facility by study staff and stored on a University of Michigan server that is password protected and secured behind firewalls. Only research staff will have access to these videos. These videos will not be shared outside the University of Michigan.

There are some reasons why people other than the researchers may need to view your study information, but they will not need to see your name or personal information. The people work for organizations that make sure our research is done safely and properly. The organizations include the University of Michigan IRB and other university offices that oversee research and the federal Office for Human Research Protections.

### **Special Protections**

This research holds a Certificate of Confidentiality from the National Institutes of Health.

This means that we cannot be forced to disclose any research information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, except as described below.

We may disclose your information for any purpose to which you have consented, as described in this informed consent document. This includes:

- 1. If you share information about future criminal conduct.
- 2. If you share any information that suggests that you may be an immediate harm to yourself or others.
- 3. If you share information about alleged or suspected child or elder abuse. However, we will not ask you questions on these topics, so you should protect your own privacy and not reveal this information.

Please note that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then we will not use the Certificate to withhold that information.

More detailed information about Certificates may be found at the NIH CoC webpage: <a href="https://humansubjects.nih.gov/coc/index">https://humansubjects.nih.gov/coc/index</a>

# What will happen to the information we collect about you after the study is over?

We plan to share the results of this study with the public. We will store your data to use for future research studies; this will include the video recordings. Your name and any other

identifying information will be secured and stored separately from your research data at the School of Social Work. Only Dr. Smith, the Principal Investigator and study team members, will have access to information that could identify you. Research data may be shared with other investigators but will never contain any information that could identify you. We will not share video recordings. De-identified data will be archived at the National Archive of Criminal Justice Data (NACJD).

There is no plan to provide you with any financial benefits from commercial products derived from the data.

#### **Voluntary Nature of the Study**

Participating in this study is completely voluntary. It is completely up to you whether you want to be in the study. Even if you say yes, you may change your mind and stop at any time. You may also choose to not answer a question for any reason. If you withdraw from the research, we will keep the data that has already been collected and continue to use it.

If you choose not to participate, this choice will not affect your relationship with the village or teachers. It will not have any impact on your treatment at the village, release, or parole status. Although your data will not be shared with correctional officials, MDOC staff could still overhear what is said and know who participates.

# **Contact Information for the Study Team**

If you have questions about this research, including questions about participating, you may contact **Dr. Matthew Smith** at <a href="mattjsmi@umich.edu">mattjsmi@umich.edu</a> or (734) 764-9322. You may also email smithlab@umich.edu.

# Contact Information for Questions about Your Rights as a Research Participant

If you have questions about your rights as a research participant, or wish to obtain information, ask questions or discuss any concerns about this study with someone other than the researcher(s), please contact the:

University of Michigan Health Sciences and Behavioral Sciences Institutional Review Board 2800 Plymouth Road

Building 520, Room 1169 Ann Arbor, MI 48109-2800

Phone: (734) 936-0933 or toll free, (866) 936-0933

Email: irbhsbs@umich.edu

#### Consent

By saying yes, you are agreeing to be in the study. We will give you a copy of this document for your records. We will keep one copy with the study records. Be sure that we have answered any questions you have about the study and you understand what you are asked to do. You may contact the researcher or the study staff if you think of a question later.

I agree to participate in the study. I understand that this means I will be audio and video recorded during the practice interview session. I understand that MDOC will provide my contact information to the research team in order to be contacted for the 6-month and 12-month follow-up survey. I understand that MDOC may also share other information about me, such as my employment status and villager status.

I understand that if I share information about future criminal conduct, if I share any information that suggests I may be an immediate harm to myself or others, or if I share information about alleged or suspected child or elder abuse, the researchers will report this information to MDOC.

Consent to be contacted for Participation in Future Research (optional)

I agree to be contacted for participation in other future research that may or may not be related to the topics of this specific project.